CLINICAL TRIAL: NCT06931041
Title: Comparing Efficacy of Autologous Serum Eye Drops With and Without Insulin in Autoimmune Dry Eye: A Randomized Clinical Trial
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Instituto de Oftalmología Fundación Conde de Valenciana (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CEI-2023/10/04
Record Dates: First submitted 2025-04-09; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Dry Eye; Sjogren Syndrome
Keywords: Dry eye; Sjogren Syndrome; Insulin; Autologous Serum
MeSH Terms: conditions — Dry Eye Syndromes; Sjogren's Syndrome; Insulin Resistance | interventions — Insulin Lispro

STUDY DESIGN:
Intervention Model Description: A randomized, single-blinded clinical trial will include patients aged 18 years and older who are diagnosed with moderate to severe DED associated with primary (PSS) or secondary (SSS) Sjögren's Syndrome. Both groups will receive ASED at a concentration of 30%. In group 2, 1 UI/ml of insulin will be added to the ASED formulation. The dosage will consist of one drop every 6 hours for 30 days in both groups. The following parameters will be evaluated at baseline (day 0), day 10, and day 30 of treatment: best corrected visual acuity (BCVA), ocular surface staining (Van-Bijsterveld score), Schirmer test, non-invasive tear break-up time (NITBUT), tear meniscus height (TMH), bulbar conjunctival hyperemia (BCH), and Ocular Surface Disease Index (OSDI) score. Statistical analysis will be performed using ANOVA for time/group comparisons with STATA 18.0 software.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Insulin (Active Comparator): 1 UI/ml of insulin added to the autologous serum formulation.
  Interventions: Drug: insulin lispro; Other: Autologous serum
- Sham (Sham Comparator): Autologous Serum without insulin.
  Interventions: Other: Autologous serum

INTERVENTIONS:
Drug: insulin lispro — 1 UI/ml of insulin added to the autologous serum formulation.
  Arms: Insulin
Other: Autologous serum — Autologous Serum

SUMMARY:
Introduction:

Dry Eye Disease (DED) of autoimmune origin is often severe and resistant to conventional treatments, necessitating alternative therapeutic options. Autologous Serum Eye Drops (ASED) have gained recognition for their biochemical and biomechanical properties, which closely mimic those of human tears. These properties make ASED an effective treatment for DED. Furthermore, topical insulin has demonstrated anti-inflammatory effects and promotes epithelial cell proliferation, differentiation, and migration, all of which contribute to maintaining ocular surface stability. As a result, insulin may serve as a valuable adjunct in treating moderate to severe autoimmune DED.

Purpose:

This study aims to assess and compare the effectiveness of autologous serum eye drops (group 1) and autologous serum eye drops combined with insulin (group 2) in improving the clinical signs and symptoms of moderate to severe DED in patients with autoimmune diseases, particularly those with Sjögren's Syndrome.

DETAILED DESCRIPTION:
Introduction:

Dry Eye Disease (DED) of autoimmune origin is often severe and resistant to conventional treatments, necessitating alternative therapeutic options. Autologous Serum Eye Drops (ASED) have gained recognition for their biochemical and biomechanical properties, which closely mimic those of human tears. These properties make ASED an effective treatment for DED. Furthermore, topical insulin has demonstrated anti-inflammatory effects and promotes epithelial cell proliferation, differentiation, and migration, all of which contribute to maintaining ocular surface stability. As a result, insulin may serve as a valuable adjunct in treating moderate to severe autoimmune DED.

Purpose:

This study aims to assess and compare the effectiveness of autologous serum eye drops (group 1) and autologous serum eye drops combined with insulin (group 2) in improving the clinical signs and symptoms of moderate to severe DED in patients with autoimmune diseases, particularly those with Sjögren's Syndrome.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria included men and women aged 18 years or older with a diagnosis of primary[ and secondary SS confirmed by a rheumatologist using the 2016 ACR-EULAR diagnostic criteria, and moderate to severe DED. Moderate to severe DED was classified using the following standardized parameters: Ocular Surface Disease Index (OSDI) ≥ 23 points, ocular surface staining according to the Van Bijsterveld score ≥ 4 points, non-invasive tear break-up time (NITBUT) ≤ 7 seconds, and tear meniscus height (TMH) ≤ 0.3 mm, measured with the Keratograph 5M (Oculus, Wetzlar, Germany). Participants were required to be willing to comply with the study protocol and follow-up schedule.

Exclusion Criteria:

* Exclusion criteria included participation in another clinical trial in the preceding three weeks, topical use of aminoglycoside antibiotics, therapeutic contact lens use, known hypersensitivity to any component of the study medications, active ocular infection, ocular surgery or trauma within three months, or any abnormality compromising corneal integrity. Additionally, patients with a history of corneal transplantation, pregnancy or lactation, or planned pregnancy were excluded.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2024-02-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
OSDI | From enrollment, 10 days and 30 days after starting treatment.
  Ocular Surface Disease Index

SECONDARY OUTCOMES:
Ocular surface staining (Van-Bijsterveld score) | From enrollment, 10 days and 30 days after starting treatment.
Schirmer test | From enrollment, 10 days and 30 days after starting treatment.
non-invasive tear break-up time (NITBUT) | From enrollment, 10 days and 30 days after starting treatment.
Tear meniscus height (TMH) | From enrollment, 10 days and 30 days after starting treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto de Oftalmologia Conde de Valenciana IAP, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: Undecided